CLINICAL TRIAL: NCT04392518
Title: Is Telerehabilitation as Effective as the Traditional Hospital-based Rehabilitation in Patients With Proximal Muscle Weakness? - A Randomized Controlled Study
Brief Title: Telerehabilitation in Proximal Muscle Weakness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018.150.IRB.1.017
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Telemedicine; Muscular Dystrophies; Proximal Myopathy
Keywords: telerehabilitation; telehealth; muscular dystrophy; proximal muscle weakness; spinal muscular atrophy; telemedicine
MeSH Terms: conditions — Muscular Dystrophies; Muscular Atrophy, Spinal | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There will be two group. The first group will perform the exercises in the hospital under the supervision of a physiotherapist (Group 1: Hospital based rehabilitation group) and the second group will perform the exercises at their home under remote supervision of a physiotherapist via internet connection (Group 2: Telerehabilitation group).
Who Masked: Outcomes Assessor
Masking Description: The assessor does not know the group of the patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital based rehabilitation group (Active Comparator): This group will perform the exercises in the hospital under the supervision of a physiotherapist
  Interventions: Other: exercise
- Telerehabilitation group (Active Comparator): This group will perform the exercises at their home under remote supervision of a physiotherapist via internet connection
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Breathing, posture, dynamic core stabilization, upper and lower extremity strengthening exercises.

SUMMARY:
The aim of our study is to investigate the effectiveness of two exercise programs supervised by a physiotherapist, performed in the hospital or at their home via electronic connection in a group of LGMD and SMA patients.

One exercise session will consist of breathing, posture, dynamic core stabilization, upper and lower extremity strengthening exercises. The basic exercises from each group will be performed as 1 set of 5 repetitions at the beginning and will be gradually increased according to the tolerability of the patient.

Fourteen subjects will be enrolled this randomized controlled study. Demographic characteristics, Vignos scale, Brooke scale, Barthel index, upper extremity functional index, Nottingham Health profile, short form-36, 6 minute walk test and muscle thicknesses measured by ultrasound of certain muscles will be recorded.

DETAILED DESCRIPTION:
Some neuromuscular diseases with myogenic or neurogenic origin present with proximal muscle weakness. These diseases preferentially affect muscles around shoulders and hips and hence are called limb girdle neuromuscular diseases (LG-NMD). Patients have difficulty in climbing stairs or hills, and reaching high shelves. The vast majority of these diseases are X-linked recessive, autosomal recessive or dominantly inherited muscular dystrophies and are called limb girdle muscular dystrophies (LGMD). Spinal muscular atrophy (SMA), a disease of motor neurons, is also characterized by progressive proximal muscle weakness. Although the diseases are progressive in both conditions, regular and proper doses of exercise starting from the early stages may delay the progression of muscle weakness and may prevent joint stiffness, and contractures.

The strengthening and aerobic exercise program increases overall wellness, condition and muscle strength in patients with neuromuscular diseases. The aerobic exercise program under supervision enhances oxidative capacity and muscle function without causing fatigue. Patients performing regular exercise program report an increase in their physical endurance, leg muscle strength and walking distance. Submaximal strengthening exercises combined with aerobic exercise are highly effective.

Regulation of the exercise program according to the needs of the patient is the most important step. Appropriate individualized exercises should be programmed by a physical medicine and rehabilitation physician and performed under the supervision of a physiotherapist in the hospital environment in order to be effective. Otherwise, success of rehabilitation and patient compliance might be reduced. With the development of technology, patients can perform exercises at their home under remote supervision by a physiotherapist via electronic connection. Therefore, the aim of our study is to investigate the effectiveness of two exercise programs supervised by a physiotherapist, performed in the hospital or at their home via electronic connection in a group of LGMD and SMA patients.

Fourteen consecutive patients from the Koç University Center for Muscle Diseases (KUCMD) diagnosed with LGMD or SMA are enrolled.

Patients followed by KUCMD outpatient clinic with proximal muscle weakness who held LGMD or SMA diagnoses will be evaluated by a physical medicine and rehabilitation physician. Demographic characteristics, Vignos scale, Brooke scale, Barthel index, upper extremity functional index, Nottingham Health profile, short form-36, 6 minute walk test and muscle thicknesses measured by ultrasound of certain muscles will be recorded. Patients will be randomized into two groups.

The first group will perform the exercises in the hospital under the supervision of a physiotherapist (Group 1: Hospital based rehabilitation group) and the second group will perform the exercises at their home under remote supervision of a physiotherapist via internet connection (Group 2: Telerehabilitation group). The exercise program will be administered 3 times in a week for 10 weeks. Patients will be examined by a blinded neurologist and functional assessments and ultrasonographic evaluations will be performed by a blinded physical medicine and rehabilitation physician before and after the rehabilitation program and at the 6th and 12th months following the completion of the rehabilitation.

One exercise session will consist of breathing, posture, dynamic core stabilization, upper and lower extremity strengthening exercises. The basic exercises from each group will be performed as 1 set of 5 repetitions at the beginning and will be gradually increased according to the tolerability of the patient. If the patient has difficulty performing the basic exercises, modifications of the relevant exercise will be applied.

ELIGIBILITY:
Inclusion Criteria:

* To be older than 18 years
* To have proximal muscle weakness with a diagnosis of LGMD of any kind and SMA
* To have ability to walk independently

Exclusion Criteria:

* history of cervical and lumbar radiculopathy
* history of cerebrovascular disease
* history of spinal cord injury

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | 6 months
  This is a field test evaluating submaximal aerobic capacity. The individuals are asked to walk as far as possible in a 30-meter corridor in 6 minutes. The technical standards are defined by European Respiratory Society and American Thoracic Society. Six minute walking distance will be recorded. Higher walking distance shows better outcome.

SECONDARY OUTCOMES:
Vignos scale | 6 months
  Vignos scale evaluates the functionality of the lower extremity and walking ability. This scale evaluates the patient's ability to standup from the chair, as well as to walk assisted with a long leg device in patients who can't walk without help. 1 indicates the best condition, 10 indicates the worst.
Brooke scale | 6 months
  Brooke scale evaluates the functionality of the upper extremity and hand skills ranging between 1- 6. 1 indicates the best condition, 6 indicates the worst.
Barthel index | 6 months
  Barthel index is a scale including ten items to assess functional disability. It is used to measure the performance of the individuals in daily life activities and the degree of care the patient needs in daily activities. 4. Total score is obtained by summing scores of 10 items. 0 indicates the worst, 100 indicates the best results.
Nottingham health profile | 6 months
  Nottingham health profile is a self-reported quality-of-life questionnaire. It consists of 38 items and evaluates 6 dimensions related to general health: energy, pain, emotional reactions, sleep, social isolation and physical activity. It is scored between 0-100 separately for each section. 0 indicates the best condition, 100 indicates the worst. The sum of the sub-scores gives the total Nottingham Health Profile score.
The upper extremity functional index | 6 months
  The upper extremity functional index. It consists of 20 items: each item is scored between 0 (extreme difficulty/inability to perform) and 4 (no difficulty) depending on the ability to perform specific activities. Total score is obtained by summing scores of 20 items. 0 indicates the worst, 80 indicates the best functional status.
Short form - 36 | 6 months
  Short form - 36 measures health related quality of life. It is a self-reported survey that evaluates individual health status with eight parameters consisting of physical function, pain, role limitations attributed to physical problems, role limitations attributed to emotional problems, mental health, social functioning, energy/ vitality, general health perception. There is not a summary score, each section is scored between 0-100, 0 indicates the worst condition, 100 indicates the best.
Muscle size and quality | 6 months
  All ultrasound evaluations will be performed using a MyLab Class C ultrasonic imaging system equipped with a 4-13-MHZ linear-array or 55 mm convex array according to the depth of the muscle. No compression to the skin will be applied. Evaluations will be performed by the same physiatrist who is blinded to the allocation groups. Measurements will be performed on the most affected side. Muscles assessed are supraspinatus, deltoid, biseps brachi for upper extremity; transversus abdominis, internal and external oblique for trunk; gluteus medius, quadriceps (rectus femoris, vastus intermedius, vastus lateralis, vastus medialis), medial gastrocnemius and hamstring muscles (semimembranosus, semitendinosus, biceps femoris) for the lower extremity. Qualitative analysis of all muscles will be performed using Heckmatt scale based on muscle echogenicity, grade 1 indicates normal, grade 4 the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Piraye Oflazer, Prof, Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was not planned to share individual participant data

REFERENCES:
- [Result] Vissing J. Limb girdle muscular dystrophies: classification, clinical spectrum and emerging therapies. Curr Opin Neurol. 2016 Oct;29(5):635-41. doi: 10.1097/WCO.0000000000000375. PMID 27490667
- [Result] Siciliano G, Simoncini C, Giannotti S, Zampa V, Angelini C, Ricci G. Muscle exercise in limb girdle muscular dystrophies: pitfall and advantages. Acta Myol. 2015 May;34(1):3-8. PMID 26155063
- [Result] Narayanaswami P, Weiss M, Selcen D, David W, Raynor E, Carter G, Wicklund M, Barohn RJ, Ensrud E, Griggs RC, Gronseth G, Amato AA; Guideline Development Subcommittee of the American Academy of Neurology; Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Evidence-based guideline summary: diagnosis and treatment of limb-girdle and distal dystrophies [RETIRED]: report of the guideline development subcommittee of the American Academy of Neurology and the practice issues review panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Neurology. 2014 Oct 14;83(16):1453-63. doi: 10.1212/WNL.0000000000000892. PMID 25313375
- [Result] Berthelsen MP, Husu E, Christensen SB, Prahm KP, Vissing J, Jensen BR. Anti-gravity training improves walking capacity and postural balance in patients with muscular dystrophy. Neuromuscul Disord. 2014 Jun;24(6):492-8. doi: 10.1016/j.nmd.2014.03.001. Epub 2014 Mar 12. PMID 24684860
- [Result] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Result] VIGNOS PJ Jr, SPENCER GE Jr, ARCHIBALD KC. Management of progressive muscular dystrophy in childhood. JAMA. 1963 Apr 13;184:89-96. doi: 10.1001/jama.1963.03700150043007. No abstract available. PMID 13997180
- [Result] Brooke MH, Griggs RC, Mendell JR, Fenichel GM, Shumate JB, Pellegrino RJ. Clinical trial in Duchenne dystrophy. I. The design of the protocol. Muscle Nerve. 1981 May-Jun;4(3):186-97. doi: 10.1002/mus.880040304. No abstract available. PMID 7017401
- [Result] Collin C, Wade DT, Davies S, Horne V. The Barthel ADL Index: a reliability study. Int Disabil Stud. 1988;10(2):61-3. doi: 10.3109/09638288809164103. PMID 3403500
- [Result] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Result] Aytar A, Yuruk ZO, Tuzun EH, Baltaci G, Karatas M, Eker L. The Upper Extremity Functional Index (UEFI): cross-cultural adaptation, reliability, and validity of the Turkish version. J Back Musculoskelet Rehabil. 2015;28(3):489-95. doi: 10.3233/BMR-140545. PMID 25322741
- [Result] Demiral Y, Ergor G, Unal B, Semin S, Akvardar Y, Kivircik B, Alptekin K. Normative data and discriminative properties of short form 36 (SF-36) in Turkish urban population. BMC Public Health. 2006 Oct 9;6:247. doi: 10.1186/1471-2458-6-247. PMID 17029646
- [Result] Ware JE: Scoring the SF-36. SF-36 Health Survey: Manual and Interpretation Guide 1993
- [Result] Heckmatt JZ, Leeman S, Dubowitz V. Ultrasound imaging in the diagnosis of muscle disease. J Pediatr. 1982 Nov;101(5):656-60. doi: 10.1016/s0022-3476(82)80286-2. PMID 7131136
- [Result] Cho J, Lee K, Kim M, Hahn J, Lee W. The Effects of Double Oscillation Exercise Combined with Elastic Band Exercise on Scapular Stabilizing Muscle Strength and Thickness in Healthy Young Individuals: A Randomized Controlled Pilot Trial. J Sports Sci Med. 2018 Mar 1;17(1):7-16. eCollection 2018 Mar. PMID 29535573
- [Result] Jenkins ND, Miller JM, Buckner SL, Cochrane KC, Bergstrom HC, Hill EC, Smith CM, Housh TJ, Cramer JT. Test-Retest Reliability of Single Transverse versus Panoramic Ultrasound Imaging for Muscle Size and Echo Intensity of the Biceps Brachii. Ultrasound Med Biol. 2015 Jun;41(6):1584-91. doi: 10.1016/j.ultrasmedbio.2015.01.017. Epub 2015 Mar 3. PMID 25746907
- [Result] Gnat R, Saulicz E, Miadowicz B. Reliability of real-time ultrasound measurement of transversus abdominis thickness in healthy trained subjects. Eur Spine J. 2012 Aug;21(8):1508-15. doi: 10.1007/s00586-012-2184-4. Epub 2012 Feb 12. PMID 22327252
- [Result] Whittaker JL, Emery CA. Sonographic measures of the gluteus medius, gluteus minimus, and vastus medialis muscles. J Orthop Sports Phys Ther. 2014 Aug;44(8):627-32. doi: 10.2519/jospt.2014.5315. Epub 2014 Jul 16. PMID 25029916
- [Result] Strasser EM, Draskovits T, Praschak M, Quittan M, Graf A. Association between ultrasound measurements of muscle thickness, pennation angle, echogenicity and skeletal muscle strength in the elderly. Age (Dordr). 2013 Dec;35(6):2377-88. doi: 10.1007/s11357-013-9517-z. Epub 2013 Mar 2. PMID 23456136
- [Result] Balius R, Pedret C, Iriarte I, Saiz R, Cerezal L. Sonographic landmarks in hamstring muscles. Skeletal Radiol. 2019 Nov;48(11):1675-1683. doi: 10.1007/s00256-019-03208-x. Epub 2019 Apr 17. PMID 30997529
- [Result] Kuyumcu ME, Halil M, Kara O, Cuni B, Caglayan G, Guven S, Yesil Y, Arik G, Yavuz BB, Cankurtaran M, Ozcakar L. Ultrasonographic evaluation of the calf muscle mass and architecture in elderly patients with and without sarcopenia. Arch Gerontol Geriatr. 2016 Jul-Aug;65:218-24. doi: 10.1016/j.archger.2016.04.004. Epub 2016 Apr 14. PMID 27107379